CLINICAL TRIAL: NCT03357562
Title: MR Imaging of Lung in the Follow-up Assessment of Cystic Fibrosis
Acronym: CFMR-lung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2016/28
Record Dates: First submitted 2017-11-15; First posted 2017-11-30 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CT; MRI; radiation dose; contrast agent
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung MRI (Experimental): lung MRI without contrast injection
  Interventions: Device: lung MRI

INTERVENTIONS:
Device: lung MRI — lung MRI without contrast injection

SUMMARY:
The aim of the study is to assess the diagnostic sensitivity of MRI to detect changes in Helbich-Bhalla scoring over time in patients with cystic fibrosis

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is caused by the cystic fibrosis transmembrane conductance regulator (CFTR) gene mutation and represents one of the most frequent and lethal inherited disease in Caucasian. However, thanks to better treatments that slow down the progression of pulmonary disease, the median life expectancy has reached 41 years and there are nowadays more CF patients older than 18-year-old than younger. Chronic lung disease is the main manifestation and represents more than 90% of CF morbidity and mortality. However, there is a need for biomarkers more sensitive than clinical and functional findings for a personalized management of patients. Computed tomography (CT), owing to its high spatial resolution and contrast, is the standard of reference in imaging for depicting lung structural alterations. But CT is an ionizing technique, rising concern in cancer risk associated to cumulated radiation dose. To date, Magnetic Resonance Imaging (MRI) is a radiation-free technique which has been demonstrated to add meaningful functional information that cannot be reached using CT. Recent advances in 3-dimensional ultra-short echo time (3D-UTE) imaging have been shown promising to improve lung MR imaging quality. A clear delineation between airway wall and lumen was obtained, thanks to submillimeter voxel size, enabling readers to estimate both bronchial thickening and dilatation with very good concordance with CT, independently from the magnitude of score. The combination of pulse sequence may rather benefit from the potential of MRI to get more complete insight into inflammatory processes by combining several contrasts, as compared to other ionizing methods. Novel MR methods have been shown promising in assessing lung changes with high resolution and therefore could be proposed instead of CT for radiation- free repeated, life-long follow-up

ELIGIBILITY:
Inclusion Criteria:

* male or female children (age ≥ 8 y.o) and adult patient with a diagnosis of cystic fibrosis provided by genetic and swear test older than 8 years. Subgroups of patients will be defined according to:

  * age: younger or older 18y.o. We expect around 50% in different subgroups. In case of, we reach 50% in one of these groups, patient recruitment will continue for both groups until the expected number of patients in the study is reached.
  * brand name of magnet: Siemens, General Electric or Philips
* new drugs use: association Ivacaftor/lumicaftor (OrkambiØ) or Ivacaftor only (Kalydeco Ø) ) We expect approximately 20% to 50% of patients treated
* Informed consent provided to the patient or/and to legal representative for adults and to parents for the children
* Patient concerned by articles L 1121-6, L 1121-7, and L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent) if the expected benefit for such persons justifies the foreseeable risk incurred

Exclusion Criteria:

* patients without any social security or health insurance
* pregnant women
* Patients with previous pulmonary transplantation or planned for transplantation in the year following inclusion
* MRI contraindications:

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of MRI to detect lung changes | Month 36
  deterioration or improvement measured by the Helbich-Bhalla scoring with CT as gold standard

SECONDARY OUTCOMES:
Sensitivity of MRI to Helbich-Bhalla scoring change | Month 0 and Month 36
  Sensitivity of MRI to Helbich-Bhalla scoring change in various subgroups of patients according to age, centers and MR scan manufacturers, and new treatment drug use (Ivacaftor/lumicaftor: Orkambi Ø or Ivacaftor : Kalydeco Ø ) from CT and MR examinations
CT / MR concordance | Month 0 and Month 36
  Concordance between CT and MR in amplitude of Helbich-Bhalla scoring variations at M0 and M36
Sensitivity of the 3D-UTE MR sequence | Month 0 and Month 36
  Sensitivity of the 3D-UTE MR sequence alone to detect change in Helbich-Bhalla scoring as compared to CT performed at M0 and M36
Imaging quality of the 3D-UTE MR | Month 0, Month 12, Month 24 and Month 36
  using a likert scale
Correlation between a specific Helbich-Bhalla MR score and the amplitude of change | Month 0 and Month 36
  Correlation between a specific Helbich-Bhalla MR score with clinical and functional data, and concordance with the amplitude of change between M0 and M36
Accuracy of a lung MR protocol | Month 0 and Month 36
  Accuracy of a lung MR protocol including T1-weighted and T2-weighted sequences to diagnose allergic broncho-pulmonary aspergillosis (ABPA) in CF patients
Reproducibility in detecting lung structural abnormality | Month 0 and Month 36
  MR and CT reproducibility in detecting lung structural abnormality at the segmental level
Reproducibility in overall Helbich-Bhalla scoring | Month 0 and Month 36
  MR and CT reproducibility in overall Helbich-Bhalla scoring
Correlations between Helbich-Bhalla scoring and clinical questionnaire | Month 0 and Month 36
  Correlations between Helbich-Bhalla scoring measured with MRI and CT and clinical questionnaire
Correlations between Helbich-Bhalla scoring and exacerbation rate | Month 0 and Month 36
  Correlations between Helbich-Bhalla scoring measured with MRI and CT and exacerbation rate
Correlations between Helbich-Bhalla scoring and clinical pulmonary functional test | Month 0 and Month 36
  Correlations between Helbich-Bhalla scoring measured with MRI and CT and clinical pulmonary functional test

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - University Hospital of Bordeaux, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHRU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hopital Nord, Marseille
  - Hopital Universitaire de la Timone, Marseille
  - Fondation Lenval, Nice
  - Hôpital Armand-Trousseau, Paris
  - Hôpital Necker Enfant Malades, Paris
  - CHRU Bretonneau-Tours, Tours